CLINICAL TRIAL: NCT03529825
Title: Rifaximin for Infection Prophylaxis in Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Muna Qayed, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00101158
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Microbial Colonization
Keywords: Rifaximin; Microbiome; Allogeneic hematopoietic stem cell transplantation; Blood stream infections; Acute graft versus host disease
MeSH Terms: conditions — Communicable Diseases | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Pilot, single arm prospective study with retrospective control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Experimental): Rifaximin will be administered twice a day orally or by nasogastric tube to patients undergoing allogeneic hematopoietic stem cell transplantation (HSCT).
  Interventions: Drug: Rifaximin
- Retrospective comparison cohort (No Intervention): Thirty six patients who underwent HSCT for hematologic malignancies, and received myeloablative conditioning, without prophylactic antibiotics, between 2013-2017 enrolled in the Aflac biorepository will comprise the comparison arm. Clinical data on transplant and infection characteristics is available and linked to stool microbiome samples already analyzed and described. Stored plasma and peripheral blood mononuclear cells are available for further analysis.

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be administered twice a day orally or by nasogastric tube, at a dose of 15 mg/kg divided BID with a maximum dose of 1,650 mg, day -7 to day +28 or discharge (maximum duration 36 days).
  Arms: Rifaximin

SUMMARY:
Primary purpose of the study is to see if rifaximin can improve the balance of bacteria within the gut, which has been shown to improve transplant outcomes. It will also assess whether rifaximin can reduce the risk of infection in blood/marrow transplant (BMT).

DETAILED DESCRIPTION:
This study is for patients who will be having a blood/marrow transplant (BMT) to treat leukemia, lymphoma or other cancer of the blood. The blood or marrow cells will come from another person (donor)-allogeneic BMT. Bacterial infections and acute graft versus host disease (AGVHD) are frequent complications of allogeneic BMT. Bacterial infections sometimes happen because injury to the gut during transplant allows gut bacteria to cross the injured gut barrier and get to the blood. AGVHD happens when certain white blood cells, called T-cells, in the donor cells (the graft) attack the patient's body.

Primary purpose of the study is to see if rifaximin can improve the balance of bacteria within the gut, which has been shown to improve transplant outcomes. It will also assess whether rifaximin can reduce the risk of infection in blood/marrow transplant (BMT).

ELIGIBILITY:
Inclusion Criteria:

1. Allogeneic HSCT recipients between the ages of 2 and 21 years.
2. Underlying hematologic malignancy, regardless of donor type or graft source.
3. Myeloablative conditioning regimen.

Exclusion Criteria:

1. Known hypersensitivity to rifaximin, or other rifamycin antimicrobial agents.
2. Minimally toxic conditioning regimen (e.g. low dose TBI based). Since these regimens induce minimal myelosuppression and gut injury, patients receiving them probably stand little to gain from antibiotic prophylaxis.
3. Patients with ongoing bacterial, viral or fungal active infections are not eligible for this study. Patients who remain on broad spectrum antibiotics for the treatment of a previous infection are not eligible.
4. The use of prophylactic antibiotics is not permitted.
5. Following the standard practice in blood and marrow transplantation, pregnant or breast feeding patients will be excluded

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Alterations to microbiome diversity in children treated with rifaximin compared to the historical cohort. | Period between the start of the preparative regimen and day 28 post transplant
  Composition will be assessed using 16S RNA sequencing. The Shannon index will be calculated for quantification of bacterial diversity.

SECONDARY OUTCOMES:
Rates of BSI pathogen infection/colonization frequency during the treatment period compared to the historical cohort. | Period between the start of the preparative regimen and day 28 post transplant
  Results of the GI pathogen panel, a test incorporated into routine patient care detecting DNA or RNA of 22 common viral, bacterial, and parasitic organisms, will provide a second assessment through molecular detection of the presence of common organisms associated with intestinal dysbiosis.
Transplant related mortality (TRM) | Period between the start of the preparative regimen and day 28 post transplant
  Number of deaths occurring in continuous complete remission.
Number of patients with Acute GVHD | Period between the start of the preparative regimen and day 100 post transplant
  Early onset (before day 100) acute GVHD (including all grades, and stratified by grades) will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual version 2, 2005, section 1 using the NIH consensus criteria
Number of patients with Chronic GVHD including overlap syndrome | Period between the start of the preparative regimen and year 5 post-transplant.
  Chronic GVHD including overlap syndrome, will be assessed according to the 2014 NIH consensus criteria.
Number of patients with other Infections | Period between the start of the preparative regimen and day 28 post transplant
  Other Infections will be defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures
Number of patients with relapse free survival at 1 year | Period between the start of the preparative regimen and year 1 post-transplant.
  Survival without relapse of underlying malignancy.
Overall number of patients survived at 1 year | Period between the start of the preparative regimen and year 1 post-transplant.
  Survival with or without relapse of underlying malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Qayed, MD MSc, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States